CLINICAL TRIAL: NCT00012818
Title: Efficacy and Cost Effectiveness of Relaxation and Response to CHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IIR 99-241
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: relaxation technique; Behavioral: educational program

INTERVENTIONS:
Behavioral: relaxation technique
Behavioral: educational program

SUMMARY:
Despite the development of significant pharmaceutical treatments, morbidity and mortality of chronic heart failure (CHF) patients remain high, patients� quality of life is poor, and their health care utilization is heavy. It is therefore important to find a cost effective non-pharmaceutical treatment to help CHF patients manage the disease. The relaxation response has been found to be effective in managing CHF-related conditions. With its favorable physiological changes, the relaxation response is likely to benefit CHF patients.

DETAILED DESCRIPTION:
Background:

Despite the development of significant pharmaceutical treatments, morbidity and mortality of chronic heart failure (CHF) patients remain high, patients� quality of life is poor, and their health care utilization is heavy. It is therefore important to find a cost effective non-pharmaceutical treatment to help CHF patients manage the disease. The relaxation response has been found to be effective in managing CHF-related conditions. With its favorable physiological changes, the relaxation response is likely to benefit CHF patients.

Objectives:

1. To evaluate the effects of a 15-week relaxation response intervention program on improving functional capacity and health-related quality of life as compared with an ongoing 15-week educational program for cardiac disease management, and a control group of usual cardiac care; 2. To identify the costs of conducting the intervention and the cardiac care education and the costs associated with cardiac care services; and to compare cost among three study groups.

Methods:

This is a single-blind three-armed randomized trial in CHF patients who receive care at the Boston VA Medical Center. Enrolled patients are randomly assigned, with equal numbers, to one of the three study groups. Outcomes include cardiac functional capacity and self-reported health-related quality of life. We also conduct a qualitative study to interview patients by phone about their experience in the study.

Status:

This project has completed the data collection phase and is in the data analysis phase.

ELIGIBILITY:
Inclusion Criteria:

CHF diagnosis, NY stage 2 or 3

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Hendricks, PhD, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA; Bei-Hung Chang, ScD, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA
Locations (1):
- Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts, United States

REFERENCES:
- [Result] Chang BH, Jones D, Hendricks A, Boehmer U, Locastro JS, Slawsky M. Relaxation response for Veterans Affairs patients with congestive heart failure: results from a qualitative study within a clinical trial. Prev Cardiol. 2004 Spring;7(2):64-70. PMID 15133373
- [Result] Chang BH, Hendricks A, Zhao Y, Rothendler JA, LoCastro JS, Slawsky MT. A relaxation response randomized trial on patients with chronic heart failure. J Cardiopulm Rehabil. 2005 May-Jun;25(3):149-57. doi: 10.1097/00008483-200505000-00005. PMID 15931018
- [Result] Chang BH, Hendricks AM, Slawsky MT, Locastro JS. Patient recruitment to a randomized clinical trial of behavioral therapy for chronic heart failure. BMC Med Res Methodol. 2004 Apr 17;4:8. doi: 10.1186/1471-2288-4-8. PMID 15090073